CLINICAL TRIAL: NCT04605419
Title: Calcium Electroporation in Patients With Barrett's Esophagus High-grade Dysplasia
Brief Title: Calcium Electroporation in Patients With Cell Changes in the Esophagus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Patrick Achiam (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor-Investigator, Michael Patrick Achiam, Consultant, MD, DMSci, Ph.D., FEBS-OG, Ass. Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEHGD-10-2020
Record Dates: First submitted 2020-10-20; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Barretts Esophagus With High Grade Dysplasia

STUDY DESIGN:
Intervention Model Description: Patients with Barrett's esophagus high-grade dysplasia will get calcium electroporation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Calcium electroporation (Experimental): Calcium chloride
  Interventions: Procedure: Calcium electroporation

INTERVENTIONS:
Procedure: Calcium electroporation — Areas with Barrett's esophagus high-grade dysplasia will get an injection of calcium chloride in submucosa through an endoscopic system before getting electroporation

SUMMARY:
The aim of this first-in-man study is to evaluate the safety of calcium electroporation used in patients with Barrett's esophagus high-grade dysplasia through an endoscopic system.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients give written informed consent. Thereafter, patient will get calcium electroporation with biopsies and digital photographs on day 0. We expect to discharge all patients same evening. Between day 3-7 an examination is followed by gastroscopy with biopsies and digital photographs. On day 14 the patients are followed in our outpatient clinic. 6 weeks after treatment the patients will undergo endoscopic mucosa resection (EMR) or endoscopic submucosa dissection (ESD) surgery and thereby the standard care of treatment for Barrett's esophagus high-grade dysplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old.
2. Histological verified Barrett's esophagus high-grade dysplasia (BE HGD)
3. Expected survival > 3 months.
4. Performance status Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) ≤ 2.
5. Platelets ≥ 50 billion/l, International Normalized Ratio (INR) < 1.5. Medical correction is allowed, e.g. correction of a high International Normalized Ratio (INR) using vitamin K.
6. Subjects must be willing and able to comply with the procedure, such as agreed follow-up visits.
7. Sexually active men and fertile women must use adequate contraception during this trial
8. Subjects must give written informed consent.

Exclusion Criteria:

1. Coagulation disorder that cannot be corrected.
2. Subjects with a clinically significant cardiac arrhythmia.
3. Concurrent treatment with an investigational medicinal product
4. Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
5. Pregnancy or lactation

A medical doctor will always be responsible for final inclusion of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Registration of treatment related side effects assessed by CTCAE V 5.0 | Day 0 to 6 weeks after treatment
  This is part of a safety evaluation and will be registered by CTCAE into Adverse Events (AE) and Serious Adverse Events (SAE)
Registration of treatment related pain through a Visual Analogue Score (VAS) | Day 0 to 6 weeks after treatment
  Second part of safety evaluation which will be registered by VAS score. The VAS score is a scale with values from 0-10, where 0 is no pain and 10 is the worst possible pain.

SECONDARY OUTCOMES:
The rate of patient's that have gained from the treatment | Day 0 to 6 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Achiam, MD., Ph.D., Principal Investigator — Rigshospitalet, Department of Surgical Gastroenterology
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark